CLINICAL TRIAL: NCT00485862
Title: Noradrenergic Augmentation of SSRI Therapy in Patients With Depression Unresponsive or Incompletely Responsive to SSRI Monotherapy
Brief Title: Combination Therapy in Patients With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6066; B4Z-MC-LYBN
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Atomoxetine Hydrochloride; Sertraline

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride
Drug: Sertraline
Drug: Placebo

SUMMARY:
The purpose of the study is to compare sertraline and atomoxetine/sertraline combination therapy in patients with persistent depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for major depression with a HAMD-17 rating scale score of at least 18 at visit 1
* Adult men or women, 18 years of age or older
* Must be able to swallow capsules
* Laboratory results must show no clinically significant abnormalities
* If suicidal ideation is present, the investigator should assess its severity and the potential need for other interventions and determine whether these are compatible with study participation

Exclusion Criteria:

* Have a documented history of Bipolar I or II disorder, or of psychosis.
* Have a history of any seizure disorder (other than febrile seizures) or patients who have taken (or are currently taking) anticonvulsants for seizure control.
* Have a history of ADHD
* Have a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions
* Are currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner which the investigator considers indicative of abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2003-06; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that augmentation of sertraline with atomoxetine for approximately 8 weeks will results in a statistically significantly greater symptom reduction in depressed patients compared with continued therapy with sertraline alone

SECONDARY OUTCOMES:
To compare the efficacy of the combination of sertraline plus atomoxetine with continued sertraline monotherapy in patients partially responsive or unresponsive to an adequate trial with sertraline monotherapy
To compare the efficacy of the combination of sertraline plus atomoxetine with continued sertraline monotherapy in the subgroup of partial responders to an adequate trial with sertraline monotherapy
To compare the efficacy of the combination of sertraline plus atomoxetine with continued sertraline monotherapy in the subgroup of nonresponders to an adequate trial with sertraline monotherapy
To compare the efficacy of the combination of sertraline plus atomoxetine with continued sertraline monotherapy in the subgroup of patients with less than a 50% reduction in baseline symptom severity after an adequate trial with sertraline monotherapy
To compare the effects of the combination of sertraline plus atomoxetine with continued sertraline monotherapy on cognition in patients with no or partial response after an adequate trail with sertraline alone
To compare the efficacy of the combination of sertraline plus atomoxetine with continued sertraline monotherapy in patients with no or partial response after an adequate trial with sertraline alone as measured by remission rates
To test the hypotheses that patients homozygous or heterozygous for the short allele of serotonin transporter will be less responsive to sertraline than patients homozygous for the long allele
To test the hypotheses that patients homozygous or heterozygous for the short allele of the serotonin transporter who have no or partial response to sertraline therapy will respond when atomoxetine is added to the treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington, United States

REFERENCES:
- [Derived] Reimherr F, Amsterdam J, Dunner D, Adler L, Zhang S, Williams D, Marchant B, Michelson D, Nierenberg A, Schatzberg A, Feldman P. Genetic polymorphisms in the treatment of depression: speculations from an augmentation study using atomoxetine. Psychiatry Res. 2010 Jan 30;175(1-2):67-73. doi: 10.1016/j.psychres.2009.01.005. Epub 2009 Dec 6. PMID 19969374
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com